CLINICAL TRIAL: NCT00736853
Title: A Phase 3 Study of JNS013 in Patients With Chronic Pain
Brief Title: An Efficacy and Safety Study of Acetaminophen Plus Tramadol Hydrochloride (JNS013) in Participants With Chronic Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR015112; JNS013-JPN-04; NCT00736853
Record Dates: First submitted 2008-08-14; First posted 2008-08-18 (Estimated); Results first posted 2013-09-26 (Estimated); Last update posted 2013-09-26 (Estimated); Status verified 2013-07

CONDITIONS: Pain
Keywords: Chronic pain; Acetoaminophen; Tramadol; Osteoarthritis of the knee; Low back pain
MeSH Terms: conditions — Pain; Chronic Pain; Osteoarthritis, Knee; Low Back Pain | interventions — Tramadol; Acetaminophen; Double-Blind Method

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tramadol Hydrochloride Plus Acetaminophen (Open-Label) (Experimental)
  Interventions: Drug: Tramadol Hydrochloride Plus Acetaminophen (Open-Label)
- Tramadol Hydrochloride Plus Acetaminophen (Double Blind) (Experimental)
  Interventions: Drug: Tramadol Hydrochloride Plus Acetaminophen (Double-Blind)
- Placebo (Double-Blind) (Placebo Comparator)
  Interventions: Drug: Placebo (Double-Blind)

INTERVENTIONS:
Drug: Tramadol Hydrochloride Plus Acetaminophen (Open-Label) — Fixed dose combination of tramadol 37.5 milligram (mg)/acetaminophen 325 mg, 1 or 2 tablets 4 times daily will be given for one week; dose level will be fixed for each participant during the second week based on analgesic efficacy and tolerability (maximum daily dose will be 8 tablets).
  Arms: Tramadol Hydrochloride Plus Acetaminophen (Open-Label)
Drug: Tramadol Hydrochloride Plus Acetaminophen (Double-Blind) — Fixed dose combination of tramadol 37.5 mg/acetaminophen 325 mg, 1 or 2 tablets (same dose [number of tablets] as that for the second week in the open-label period) will be given 4 times daily up to 4 weeks.
  Arms: Tramadol Hydrochloride Plus Acetaminophen (Double Blind)
Drug: Placebo (Double-Blind) — Matching placebo will be given up to 4 weeks.
  Arms: Placebo (Double-Blind)

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of tramadol hydrochloride plus acetaminophen (JNS013) in participants with chronic pain accompanied by osteoarthritis (a progressive and degenerative joint disease, in which the joints become painful and stiff) of the knee or low back pain (acute or chronic pain in the lumbar or sacral regions) which cannot be controlled sufficiently with non-steriodal anti-inflammatory drugs (NSAIDs).

DETAILED DESCRIPTION:
This is a multi-center (when more than one hospital or medical school team work on a medical research study), double-blind (test or experiment in which neither the person giving the treatment nor the participant knows which treatment the participant is receiving), placebo-controlled (an inactive substance; a pretend treatment [with no drug in it] that is compared in a clinical trial with a drug to test if the drug has a real effect), parallel group comparison study. The total duration of the study will be 11 weeks and consists of 4 periods; a pre-observation period (4 weeks), open-label period (2 weeks), double-blind period (4 weeks) and follow-up period (1 week). Participants will receive tramadol hydrochloride plus acetaminophen tablets orally 4 times daily for 2 weeks with no less than 4-hour intervals (up to 8 tablets per day) during the open-label period and the dose will be fixed for each participant in the latter 1 week. During the double-period participants will receive tramadol hydrochloride plus acetaminophen tablets or placebo at the same dose as used for the latter 1 week of the open-label period for up to 4 weeks. Efficacy will be primarily evaluated by number of participants with insufficient pain relief after the start of double-blind period. Participant's safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants with sustention of chronic pain associated with OA or LBP for at least 3 months
* Participants whose pain cannot be controlled sufficiently with at least 14-day continuous treatment with identical oral NSAIDs at a usual maximum dose during 3 months prior to this study
* Outpatients
* Ambulatory participants without need for any supportive device or assistance during daily life

Exclusion Criteria:

* Participants with conditions for which opioids are contraindicated
* Participants with conditions for which acetaminophen is contraindicated
* Participants with history of convulsion or the possibility of convulsive seizure
* Participants with concurrent, previous, or possible alcohol dependence, drug dependence, or narcotic addiction
* Pregnant participants or those who may be pregnant, lactating mothers, and participants who wish pregnancy during the study period

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2008-06; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K. Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (20):
- Japan (20):
  - Aichi
  - Amagasaki
  - Chiba
  - Edogawa City
  - Fukuoka
  - Fukushima
  - Iruma
  - Kagoshima
  - Kawasaki
  - Kumagaya
  - Kurume
  - Meguro City
  - Minato
  - Niigata
  - Ohta-Ku
  - Okazaki
  - Sagamihara
  - Setagaya City
  - Shibuya City
  - Shinjuku-Ku

REFERENCES:
- See also: A Phase III Study of JNS013 in Patients with Chronic Pain — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=423&filename=CR015112_CSR.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Tramadol Hydrochloride and Acetaminophen (Open-Label): Fixed dose combination of tramadol 37.5 milligram (mg)/acetaminophen 325 mg, 1 or 2 tablets 4 times daily was given for one week; dose level was fixed for each participant during the second week based on analgesic efficacy and tolerability (maximum daily dose was 8 tablets).
- Tramadol Hydrochloride and Acetaminophen (Double-Blind): Fixed dose combination of tramadol 37.5 mg/acetaminophen 325 mg, 1 or 2 tablets (same dose [number of tablets] as that for the second week in the open-label period) was given 4 times daily up to 4 weeks.
- Placebo (Double-Blind): Matching placebo was given up to 4 weeks.
Period: Open-Label Period
Arm/Group | Tramadol Hydrochloride and Acetaminophen (Open-Label) | Tramadol Hydrochloride and Acetaminophen (Double-Blind) | Placebo (Double-Blind)
Started | 319 | 0 | 0
Treated | 277 | 0 | 0
Completed | 187 | 0 | 0
Not Completed | 132 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 0
Not completed — Adverse Event | 31 | 0 | 0
Not completed — Withdrawal by Subject | 16 | 0 | 0
Not completed — Started but not treated | 42 | 0 | 0
Not completed — Failed to meet the transfer criteria | 40 | 0 | 0
Not completed — Unable to attend hospital appointments | 1 | 0 | 0
Period: Double-Blind Period
Arm/Group | Tramadol Hydrochloride and Acetaminophen (Open-Label) | Tramadol Hydrochloride and Acetaminophen (Double-Blind) | Placebo (Double-Blind)
Started | 0 | 94 | 93
Completed | 0 | 70 | 45
Not Completed | 0 | 24 | 48
Not completed — Lack of Efficacy | 0 | 19 | 42
Not completed — Adverse Event | 0 | 3 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 4
Not completed — Ineligible to participate the study | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Fixed dose combination of tramadol 37.5 milligram (mg)/acetaminophen 325 mg, 1 or 2 tablets 4 times daily was given for one week; dose level was fixed for each participant during the second week based on analgesic efficacy and tolerability (maximum daily dose was 8 tablets) during the open-label period. Participants received placebo or fixed dose combination of tramadol 37.5 mg/acetaminophen 325 mg (same dose which was used in second week of open-label period) in double-blind period.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 277
Age Continuous [Mean (Standard Deviation); unit: years] — Efficacy analysis set: Participants who received at least 1 dose of study drug.
  years | 57.0 (17.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Efficacy analysis set: Participants who received at least 1 dose of study drug.
  Participants
    Female | 168
    Male | 109

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Insufficient Pain Relief After the Start of Double-Blind Period
Description: The pain relief was regarded as insufficient, if either of the following was met, a) the value of average pain intensity felt in daily living during the past 24 hours (Visual analog scale 24 [VAS24] ) on 2 consecutive days in double-blind period worsened greater than 15 millimeter (mm) compared with the average VAS24 during 3 days before the end of open-label period, b) when the participant asked for discontinuation of treatment with the study drug because of insufficient pain relief.
Time Frame: Day 28 of double-blind period
Population: Efficacy analysis set included participants who received at least one dose of the study drug.
Measure: Number; unit: number of participants
Arm/Group | Tramadol Hydrochloride and Acetaminophen (Double-Blind) | Placebo (Double-Blind)
Number analyzed (Participants) | 94 | 93
number of participants | 20 | 43
Statistical Analysis 1: Comparison: Tramadol Hydrochloride and Acetaminophen (Double-Blind) vs Placebo (Double-Blind); Test type: Superiority or Other; p = 0.0001, Log Rank; Stratified Log-rank test with the target disease as the stratification factor; Hazard Ratio (HR) = 0.377, 95% CI 2-sided [0.221 to 0.641]

2. Secondary Outcome: Change in the Visual Analog Scale for the Last 24 Hours (VAS24) Value at the Start of the Double-Blind Period From the Baseline Value at the Start of the Open-Label Period
Description: Pain over the last 24 hours was assessed by using VAS score ranges from 0 mm=no pain to 100 mm=worst possible pain. An increase in score from Baseline represented disease progression and decrease represented improvement.
Time Frame: Day 1 of open-label period and Day 1 of double-blind period
Population: Efficacy analysis set included participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tramadol Hydrochloride and Acetaminophen (Open-Label)
Number analyzed (Participants) | 277
mm
  Day 1 of open-label period | 66.27 (13.69)
  Change at Day 1 of double-blind period | -28.17 (21.16)

3. Secondary Outcome: Change in the VAS24 Value From the Baseline at the Final Time Point of the Double-Blind Period
Description: as for outcome 2
Time Frame: Day 1 and Day 28 of double-blind period
Population: Efficacy analysis set included participants who received at least one dose of the study drug.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tramadol Hydrochloride and Acetaminophen (Double-Blind) | Placebo (Double-Blind)
Number analyzed (Participants) | 94 | 93
mm
  Day 1 | 30.33 (17.47) | 31.18 (16.59)
  Change at Day 28 | -0.67 (18.14) | 6.21 (22.50)

4. Secondary Outcome: Mean Pain Intensity (PI) Score During Open-Label Period
Description: PI was evaluated on a 4-stage scale with a score ranging from 0 to 3, wherein 0=no pain and 3=severe pain.
Time Frame: Pre-dose and post-dose at 2 hours, 4 hours on Day 1, and Day 8 of open-label period
Population: Efficacy analysis set included participants who received at least one dose of study drug. Here 'n' signifies number of participants evaluable for this outcome measure at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tramadol Hydrochloride and Acetaminophen (Open-Label)
Number analyzed (Participants) | 277
units on a scale
  Day 1; Pre-dose (n=275) | 1.7 (0.56)
  Day 1; 2 hours after dosing (n=274) | 1.2 (0.62)
  Day 1; 4 hours after dosing (n=274) | 1.1 (0.65)
  Day 8; Pre-dose (n=219) | 1.2 (0.43)
  Day 8; 2 hours after dosing (n=219) | 1.0 (0.49)
  Day 8; 4 hours after dosing (n=219) | 0.9 (0.55)

5. Secondary Outcome: Mean PI Score During Double-Blind Period
Description: The PI was evaluated on a 4-stage scale with a score ranging from 0 to 3, wherein 0=no pain and 3=severe pain.
Time Frame: Pre-dose and post-dose at 2 hours, 4 hours on Day 1, 8, 15, 22 and 28 of double-blind period
Population: Efficacy analysis set included participants who received at least one dose of the study drug. Here 'n' signifies number of participants evaluable at each time point for each arm respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tramadol Hydrochloride and Acetaminophen (Double-Blind) | Placebo (Double-Blind)
Number analyzed (Participants) | 94 | 93
units on a scale
  Day 1; Pre-dose (n=84, 89) | 1.2 (0.37) | 1.2 (0.37)
  Day 1; 2 hours after dosing (n=84, 89) | 1.0 (0.44) | 1.1 (0.43)
  Day 1; 4 hours after dosing (n=84, 89) | 1.0 (0.49) | 1.1 (0.47)
  Day 8; Pre-dose (n=74, 48) | 1.2 (0.39) | 1.2 (0.42)
  Day 8; 2 hours after dosing (n=74, 48) | 1.0 (0.47) | 1.1 (0.58)
  Day 8; 4 hours after dosing (n=74, 48) | 0.9 (0.51) | 1.1 (0.43)
  Day 15; Pre-dose (n=67, 41) | 1.1 (0.33) | 1.1 (0.33)
  Day 15; 2 hours after dosing (n=67, 41) | 1.0 (0.46) | 1.0 (0.50)
  Day 15; 4 hours after dosing (n=67, 41) | 0.8 (0.51) | 0.9 (0.52)
  Day 22; Pre-dose (n=63, 40) | 1.1 (0.30) | 1.2 (0.38)
  Day 22, 2 hours after dosing (n=63, 40) | 1.0 (0.42) | 1.0 (0.50)
  Day 22; 4 hours after dosing (n=63, 40) | 0.9 (0.49) | 1.0 (0.50)
  Day 28; Pre-dose (n=72, 47) | 1.1 (0.33) | 1.2 (0.41)
  Day 28; 2 hours after dosing (n=72, 47) | 1.0 (0.44) | 1.0 (0.51)
  Day 28; 4 hours after dosing (n=72, 47) | 0.9 (0.50) | 1.0 (0.49)

6. Secondary Outcome: Mean Pain Intensity Difference (PID) During the Open-Label Period
Description: The PID was calculated as PI at pre-dose on Day 1, 8 minus PI at post-dose time point (i.e., 2 hours and 4 hours) on Day 1, 8 respectively. Baseline PI score ranges from 1=minor to 3=severe, post-baseline PI score ranges from 0=none to 3=severe. Total possible score range for PID: -2=worst to 3=best.
Time Frame: Pre-dose, and post-dose at 2 hours, 4 hours on Day 1, and Day 8 of open-label period
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tramadol Hydrochloride and Acetaminophen (Open-Label)
Number analyzed (Participants) | 277
units on a scale
  Day 1; 2 hours after dosing (n=274) | 0.4 (0.59)
  Day 1; 4 hours after dosing (n=274) | 0.5 (0.66)
  Day 8; 2 hours after dosing (n=219) | 0.2 (0.50)
  Day 8; 4 hours after dosing (n=219) | 0.3 (0.52)

7. Secondary Outcome: Mean PID During the Double-Blind Period
Description: The PID was calculated as PI at pre-dose on Day 1, 8, 15, 22, 28 minus PI at post-dose time point (i.e., 2 hours and 4 hours) on Day 1, 8, 15, 22, 28 respectively. Baseline PI score ranges from 1=minor to 3=severe, post-baseline PI score ranges from 0=none to 3=severe. Total possible score range for PID: -2=worst to 3=best.
Time Frame: Pre-dose, and post-dose at 2 hours, 4 hours on Day 1, 8, 15, 22 and 28 of double-blind period
Population: Efficacy analysis set included participants received at least one dose of the study drug. Here 'n' signifies number of participants evaluable at each time point for each arm respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tramadol Hydrochloride and Acetaminophen (Double-Blind) | Placebo (Double-Blind)
Number analyzed (Participants) | 94 | 93
units on a scale
  Day 1; 2 hours after dosing (n=84, 89) | 0.2 (0.40) | 0.1 (0.34)
  Day 1; 4 hours after dosing (n=84, 89) | 0.2 (0.49) | 0.1 (0.42)
  Day 8; 2 hours after dosing (n=74, 48) | 0.2 (0.39) | 0.1 (0.46)
  Day 8; 4 hours after dosing (n=74, 48) | 0.3 (0.50) | 0.2 (0.38)
  Day 15; 2 hours after dosing (n=67, 41) | 0.1 (0.36) | 0.2 (0.44)
  Day 15; 4 hours after dosing (n=67, 41) | 0.3 (0.49) | 0.2 (0.51)
  Day 22; 2 hours after dosing (n=63, 40) | 0.1 (0.35) | 0.2 (0.42)
  Day 22; 4 hours after dosing (n=63, 40) | 0.2 (0.42) | 0.2 (0.42)
  Day 28; 2 hours after dosing (n=72, 47) | 0.2 (0.36) | 0.2 (0.41)
  Day 28; 4 hours after dosing (n=72, 47) | 0.3 (0.44) | 0.2 (0.43)

8. Secondary Outcome: Mean Pain Relief (PAR) Score During the Open-Label Period
Description: PAR was evaluated based on 5-stage scale with a score ranging from 0 to 4, wherein, 0=no relief and 4=complete relief.
Time Frame: 2 hours, 4 hours post-dose on Day 1, and Day 8 of open-label period
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tramadol Hydrochloride and Acetaminophen (Open-Label)
Number analyzed (Participants) | 277
units on a scale
  Day 1; 2 hours after dosing (n=274) | 1.2 (0.97)
  Day 1; 4 hours after dosing (n=274) | 1.4 (1.01)
  Day 8; 2 hours after dosing (n=219) | 1.7 (1.03)
  Day 8; 4 hours after dosing (n=219) | 1.8 (1.02)

9. Secondary Outcome: Mean PAR Score During the Double-Blind Period
Description: PAR was evaluated based on 5-stage scale with a score ranging from 0 to 4, wherein, 0=no relief and 4=complete relief.
Time Frame: 2 hours, 4 hours post-dose on Day 1, 8, 15, 22 and 28 of double-blind period
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tramadol Hydrochloride and Acetaminophen (Double-Blind) | Placebo (Double-Blind)
Number analyzed (Participants) | 94 | 93
units on a scale
  Day 1; 2 hours after dosing (n=84, 89) | 1.7 (1.02) | 1.1 (1.04)
  Day 1; 4 hours after dosing (n=84, 89) | 1.8 (1.01) | 1.2 (1.00)
  Day 8; 2 hours after dosing (n=74, 48) | 1.9 (1.06) | 1.2 (1.08)
  Day 8; 4 hours after dosing (n=74, 48) | 1.9 (1.01) | 1.4 (1.05)
  Day 15; 2 hours after dosing (n=67, 41) | 2.1 (1.09) | 1.7 (1.11)
  Day 15; 4 hours after dosing (n=67, 41) | 2.1 (1.00) | 1.7 (1.06)
  Day 22; 2 hours after dosing (n=63, 40) | 2.1 (0.96) | 1.8 (1.21)
  Day 22; 4 hours after dosing (n=63, 40) | 2.2 (1.00) | 1.8 (1.26)
  Day 28; 2 hours after dosing (n=72, 47) | 2.1 (1.00) | 1.6 (1.26)
  Day 28; 4 hours after dosing (n=72, 47) | 2.1 (1.04) | 1.7 (1.29)

10. Secondary Outcome: Pain Intensity Difference and Pain Relief Scores (PRID) During the Open-Label Period
Description: The PRID is defined as sum of PID and PAR Scores for each participant at each evaluation time point (at 2 and 4 hours after the dosing). The overall possible score ranges for PRID is -2=worst to 7=best. The PID was calculated as PI at pre-dose on Day 1, 8 minus PI at post-dose time point (i.e., 2 hours and 4 hours) on Day 1, 8 respectively. Baseline PI score ranges from 1=minor to 3=severe, post-baseline PI score ranges from 0=none to 3=severe. Total possible score range for PID: -2=worst to 3=best and PAR was evaluated based on a 5-stage scale score ranges from 0=no relief and 4=complete relief.
Time Frame: 2 hours, 4 hours post-dose on Day 1, and Day 8 of open-label period
Population: Efficacy analysis set included who received at least one dose of study medication. Here 'n' signifies number of participants evaluable for each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tramadol Hydrochloride and Acetaminophen (Open-Label)
Number analyzed (Participants) | 277
units on a scale
  Day 1; 2 hours after dosing (n=274) | 1.6 (1.39)
  Day 1; 4 hours after dosing (n=274) | 1.9 (1.49)
  Day 8; 2 hours after dosing (n=219) | 1.9 (1.30)
  Day 8; 4 hours after dosing (n=219) | 2.2 (1.36)

11. Secondary Outcome: Pain Intensity Difference and Pain Relief Scores (PRID) During the Double-Blind Period
Description: The PRID is defined as sum of PID and PAR Scores for each participant at each evaluation time point (at 2 and 4 hours after the dosing). The overall possible score range for PRID is -2=worst to 7=best. The PID was calculated as PI at pre-dose on Day 1, 8, 15, 22, 28 minus PI at post-dose time point (i.e., 2 hours and 4 hours) on Day 1, 8, 15, 22, 28 respectively. Baseline PI score ranges from 1=minor to 3=severe, post-baseline PI score ranges from 0=none to 3=severe. Total possible score range for PID: -2=worst to 3=best and PAR was evaluated based on a 5-stage scale score ranges from 0=no relief and 4=complete relief.
Time Frame: 2 hours, 4 hours post-dose on Day 1, 8, 15, 22 and 28 of double-blind period
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tramadol Hydrochloride and Acetaminophen (Double-Blind) | Placebo (Double-Blind)
Number analyzed (Participants) | 94 | 93
units on a scale
  Day 1; 2 hours after dosing (n=84, 89) | 1.9 (1.20) | 1.2 (1.19)
  Day 1; 4 hours after dosing (n=84, 89) | 2.0 (1.28) | 1.2 (1.18)
  Day 8; 2 hours after dosing (n=74, 48) | 2.1 (1.23) | 1.4 (1.36)
  Day 8; 4 hours after dosing (n=74, 48) | 2.3 (1.22) | 1.6 (1.25)
  Day 15; 2 hours after dosing (n=67, 41) | 2.2 (1.29) | 1.8 (1.39)
  Day 15; 4 hours after dosing (n=67, 41) | 2.4 (1.27) | 1.9 (1.35)
  Day 22; 2 hours after dosing (n=63, 40) | 2.3 (1.10) | 2.0 (1.46)
  Day 22; 4 hours after dosing (n=63, 40) | 2.4 (1.24) | 2.1 (1.45)
  Day 28; 2 hours after dosing (n=72, 47) | 2.2 (1.14) | 1.8 (1.52)
  Day 28; 4 hours after dosing (n=72, 47) | 2.4 (1.28) | 1.9 (1.49)

12. Secondary Outcome: Sum of Pain Intensity Difference (SPID) Score During the Open-Label Period
Description: The SPID is defined as sum of the PID at 2 and 4 hours after dosing on each evaluation day. The overall possible score ranges for SPID is -4=worst to 6=best. The PID was calculated as PI at pre-dose on Day 1, 8 minus PI at post-dose time point (i.e., 2 hours and 4 hours) on Day 1, 8 respectively. Baseline PI score ranges from 1=minor to 3=severe, post-baseline PI score ranges from 0=none to 3=severe. Total possible score range for PID: -2=worst to 3=best.
Time Frame: Day 1, and Day 8 of open-label period
Population: Efficacy analysis set included participants received at least one dose of the study drug. Here 'n' signifies number of participants evaluable for this outcome measure at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tramadol Hydrochloride and Acetaminophen (Open-Label)
Number analyzed (Participants) | 277
units on a scale
  Day 1 (n=274) | 0.9 (1.17)
  Day 8 (n=219) | 0.5 (0.93)

13. Secondary Outcome: Sum of Pain Intensity Difference (SPID) Score During the Double-Blind Period
Description: The SPID is defined as sum of the PID at 2 and 4 hours after dosing on each evaluation day. The overall possible score ranges for SPID is -4=worst to 6=best. The PID was calculated as PI at pre-dose on Day 1, 8, 15, 22, 28 minus PI at post-dose time point (i.e., 2 hours and 4 hours) on Day 1, 8, 15, 22, 28 respectively. Baseline PI score ranges from 1=minor to 3=severe, post-baseline PI score ranges from 0=none to 3=severe. Total possible score range for PID: -2=worst to 3=best.
Time Frame: Day 1, 8, 15, 22 and 28 of double-blind period
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tramadol Hydrochloride and Acetaminophen (Double-Blind) | Placebo (Double-Blind)
Number analyzed (Participants) | 94 | 93
units on a scale
  Day 1 (n=84, 89) | 0.4 (0.79) | 0.1 (0.70)
  Day 8 (n=74, 48) | 0.5 (0.81) | 0.3 (0.78)
  Day 15 (n=67, 41) | 0.4 (0.76) | 0.4 (0.86)
  Day 22 (n=63, 40) | 0.4 (0.73) | 0.5 (0.78)
  Day 28 (n=72, 47) | 0.4 (0.74) | 0.4 (0.77)

14. Secondary Outcome: Total Pain Relief (TOTPAR) Score During the Open-Label Period
Description: The TOTPAR is defined as sum of PAR at 2 hours after dosing and the PAR at 4 hours after dosing on each evaluation day. Pain relief as evaluated on 5-stage scale with a score ranging from 0=no relief and 4=complete relief. Total possible score range for TOTPAR is 0=no relief to 8=complete relief.
Time Frame: Day 1 and Day 8 of open-label period
Population: Efficacy analysis set included who received at least one dose of study drug. Here 'n' signifies number of participants evaluable for each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tramadol Hydrochloride and Acetaminophen (Open-Label)
Number analyzed (Participants) | 277
units on a scale
  Day 1 (n=274) | 2.6 (1.89)
  Day 8 (n=219) | 3.5 (1.95)

15. Secondary Outcome: Total Pain Relief (TOTPAR) Score During the Double-Blind Period
Description: as for outcome 14
Time Frame: Day 1, 8, 15, 22 and 28 of double-blind period
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tramadol Hydrochloride and Acetaminophen (Double-Blind) | Placebo (Double-Blind)
Number analyzed (Participants) | 94 | 93
units on a scale
  Day 1 (n=84, 89) | 3.5 (1.97) | 2.3 (2.00)
  Day 8 (n=74, 48) | 3.8 (2.00) | 2.6 (2.05)
  Day 15 (n=67, 41) | 4.1 (2.04) | 3.3 (2.10)
  Day 22 (n=63, 40) | 4.3 (1.91) | 3.6 (2.42)
  Day 28 (n=72, 47) | 4.2 (1.99) | 3.3 (2.50)

16. Secondary Outcome: Sum of Pain Relief Combined With Pain Intensity Difference (SPRID) Score During the Open-Label Period
Description: The SPRID is defined as sum of PID and PAR Scores at 2 hours and 4 hours after the dosing on each evaluation day. The overall possible score ranges for SPRID is -4=worst to 14=best. The PID was calculated as PI at pre-dose on Day 1, 8 minus PI at post-dose time point (i.e., 2 hours and 4 hours) on Day 1, 8 respectively. Baseline PI score ranges from 1=minor to 3=severe, post-baseline PI score ranges from 0=none to 3=severe. Total possible score range for PID: -2=worst to 3=best and PAR was evaluated based on 5-stage scale with a score ranging from 0=no relief to 4=complete relief.
Time Frame: Day 1, and Day 8 of open-label period
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tramadol Hydrochloride and Acetaminophen (Open-Label)
Number analyzed (Participants) | 277
units on a scale
  Day 1 (n=274) | 3.5 (2.74)
  Day 8 (n=219) | 4.1 (2.50)

17. Secondary Outcome: Sum of Pain Relief Combined With Pain Intensity Difference (SPRID) Score During the Double-Blind Period
Description: The SPRID is defined as sum of PID and PAR Scores at 2 hours and 4 hours after the dosing on each evaluation day. The overall possible score ranges for SPRID is -4=worst to 14=best. The PID was calculated as PI at pre-dose on Day 1, 8, 15, 22, 28 minus PI at post-dose time point (i.e., 2 hours and 4 hours) on Day 1, 8, 15, 22, 28 respectively. Baseline PI score ranges from 1=minor to 3=severe, post-baseline PI score ranges from 0=none to 3=severe. Total possible score range for PID: -2=worst to 3=best and PAR was evaluated based on 5-stage scale with a score ranging from 0 to 4, wherein, 0=no relief and 4=complete relief.
Time Frame: Day 1, 8, 15, 22 and 28 of double-blind period
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tramadol Hydrochloride and Acetaminophen (Double-Blind) | Placebo (Double-Blind)
Number analyzed (Participants) | 94 | 93
units on a scale
  Day 1 (n=84, 89) | 3.9 (2.37) | 2.4 (2.30)
  Day 8 (n=74, 48) | 4.3 (2.32) | 3.0 (2.48)
  Day 15 (n=67, 41) | 4.6 (2.46) | 3.7 (2.61)
  Day 22 (n=63, 40) | 4.7 (2.27) | 4.0 (2.81)
  Day 28 (n=72, 47) | 4.6 (2.35) | 3.7 (2.90)

18. Secondary Outcome: Change From Baseline in Roland Morris Disability Questionnaire (RDQ) Total Score at Day 14 of Open-Label Period
Description: The RDQ is self-administered measure of disability caused by low back pain and consists of 24 statements. The total score ranges from 0=no disability to 24=severe disability. The higher scores indicate greater physical disability.
Time Frame: Day 1 and Day 14 of open-label period
Population: Efficacy analysis set included who received at least one dose of study drug and had the lumbago as the target disease. Here 'n' signifies number of participants evaluable for this outcome measure at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tramadol Hydrochloride and Acetaminophen (Open-Label)
Number analyzed (Participants) | 160
units on a scale
  Day 1 (n=160) | 9.1 (4.89)
  Change at Day 14 (n=126) | -2.6 (3.28)

19. Secondary Outcome: Change From Baseline in RDQ Total Score at Day 28 of Double-Blind Period
Description: as for outcome 18
Time Frame: Day 1 and Day 28 of double-blind period
Population: Efficacy analysis set included participants received at least one dose of the study drug and had the lumbago as the target disease. Here 'n' signifies number of participants evaluable at each time point for each arm respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tramadol Hydrochloride and Acetaminophen (Double-Blind) | Placebo (Double-Blind)
Number analyzed (Participants) | 55 | 57
units on a scale
  Day 1 (n=55, 57) | 6.5 (4.41) | 6.0 (4.57)
  Change at Day 28 (n=55, 57) | -0.5 (3.08) | 0.8 (3.69)

20. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Questionnaire Score at Day 14 of Open-Label Period
Description: The WOMAC questionnaire is an activity of daily living (ADL) indicator for Knee Osteoarthritis and designed to capture the elements of pain, stiffness, extent of obstruction to daily activities (EODA) and general index. The score for each element ranges from 0=better ADL to 10=worse ADL.
Time Frame: Day 1 and Day 14 of open-label period
Population: Efficacy analysis set included who received at least one dose of study drug and had the knee osteoarthritis as the target disease. Here 'n' signifies number of participants evaluable for this outcome measure at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Tramadol Hydrochloride and Acetaminophen (Open-Label): Fixed dose combination of tramadol 37.5 mg/acetaminophen 325 mg, 1 or 2 tablets (same dose [number of tablets] as that for the second week in the open-label period) was given 4 times daily up to 4 weeks.
Arm/Group | Tramadol Hydrochloride and Acetaminophen (Open-Label)
Number analyzed (Participants) | 117
units on a scale
  Day 1; Pain (n=117) | 4.4 (1.96)
  Change at Day 14; Pain (n=90) | -1.9 (1.66)
  Day 1; Stiffness (n=117) | 4.2 (2.31)
  Change at Day 14; Stiffness (n=90) | -1.5 (2.09)
  Day 1; EODA (n=117) | 3.7 (1.89)
  Change at Day 14; EODA (n=90) | -1.5 (1.38)
  Day 1; General index (n=117) | 4.1 (1.82)
  Change at Day 14; General index (n=90) | -1.7 (1.39)

21. Secondary Outcome: Change From Baseline in WOMAC Questionnaire Score at Day 28 of Double-Blind Period
Description: as for outcome 20
Time Frame: Day 1 and Day 28 of double-blind period
Population: Efficacy analysis set included who received at least one dose of study drug and had the knee osteoarthritis as the target disease. Here 'n' signifies number of participants evaluable at each time point for each arm respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tramadol Hydrochloride and Acetaminophen (Double-Blind) | Placebo (Double-Blind)
Number analyzed (Participants) | 39 | 36
units on a scale
  Day 1; Pain (n=39, 36) | 2.6 (1.46) | 2.2 (1.20)
  Change at Day 28; Pain (n=39, 36) | -0.3 (1.02) | 0.5 (1.49)
  Day 1; Stiffness (n=39, 36) | 2.7 (1.94) | 2.4 (1.72)
  Change at Day 28; Stiffness (n=39, 36) | -0.2 (1.33) | 0.2 (1.99)
  Day 1; EODA (n=39, 36) | 2.3 (1.68) | 1.9 (1.45)
  Change at Day 28; EODA (n=39, 36) | -0.5 (0.58) | 0.4 (1.30)
  Day 1; General index (n=39, 36) | 2.5 (1.48) | 2.2 (1.23)
  Change at Day 28; General index (n=39, 36) | -0.4 (0.65) | 0.4 (1.29)

22. Secondary Outcome: Change From Baseline in Short Form-36 (SF-36) Score at Day 14 of Open-Label Period
Description: The SF-36 is a survey of participant health and quality of life. It consists of 8 sub-scales, which are the weighted sums of the questions in their section. The 8 sub-scales are: physical functioning, role-physical, role-emotional, general health, social functioning, bodily pain, vitality, mental health. Each item is scored on a scale ranging from 0-100. Higher score defines a more favorable health status or a better mental status.
Time Frame: Day 1 and Day 14 of open-label period
Population: Efficacy analysis set included who received at least one dose of study drug. Here 'n' signifies number of participants evaluable for this outcome measure at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tramadol Hydrochloride and Acetaminophen (Open-Label)
Number analyzed (Participants) | 277
units on a scale
  Day 1; Physical functioning (n=277) | 34.3 (15.23)
  Change at Day 14; Physical functioning (n=216) | 3.9 (10.39)
  Day 1; Role-physical (n=216) | 37.0 (13.62)
  Change at Day 14; Role-physical (n=216) | 4.3 (11.10)
  Day 1; Bodily pain (n=277) | 34.8 (6.59)
  Change at Day 14; Bodily pain (n=216) | 5.4 (7.04)
  Day 1; General health (n=277) | 45.4 (9.01)
  Change at Day 14; General health (n=216) | 2.7 (6.31)
  Day 1; Vitality (n=277) | 45.1 (9.43)
  Change at Day 14; Vitality (n=216) | 2.3 (8.10)
  Day 1; Social functioning (n=277) | 43.5 (12.48)
  Change at Day 14; Social functioning (n=277) | 2.0 (10.76)
  Day 1; Role-emotional (n=277) | 43.2 (12.95)
  Change at Day 14; Role-emotional (n=216) | 2.5 (11.36)
  Day 1; Mental health (n=277) | 46.8 (9.69)
  Change at Day 14; Mental health (n=216) | 2.8 (8.59)

23. Secondary Outcome: Change From Baseline in SF-36 at Day 28 of Double-Blind Period
Description: as for outcome 22
Time Frame: Day 1 and Day 28 of double-blind period
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tramadol Hydrochloride and Acetaminophen (Double-Blind) | Placebo (Double-Blind)
Number analyzed (Participants) | 94 | 93
units on a scale
  Day 1; Physical functioning (n=94,93) | 39.0 (12.28) | 39.7 (13.36)
  Change at Day 28; Physical functioning (n=94,93) | 1.1 (8.49) | -1.6 (10.03)
  Day 1; Role-physical (n=94,93) | 40.5 (12.84) | 41.8 (12.24)
  Change at Day 28; Role-physical (n=94,93) | 0.8 (11.87) | -0.6 (9.54)
  Day 1; Bodily pain (n=94,93) | 41.0 (7.68) | 39.3 (7.27)
  Change at Day 28; Bodily pain (n=94,93) | 2.4 (7.24) | 0.3 (7.77)
  Day 1; General health (n=94,93) | 49.1 (9.23) | 48.0 (9.33)
  Change at Day 28; General health (n=94,93) | 0.4 (7.11) | -1.2 (5.97)
  Day 1; Vitality (n=94,93) | 47.3 (9.58) | 47.4 (8.49)
  Change at Day 28; Vitality (n=94,93) | 3.1 (7.40) | 0.1 (7.51)
  Day 1; Social functioning (n=94,93) | 46.4 (12.68) | 45.7 (11.48)
  Change at Day 28; Social functioning (n=94,93) | 1.6 (11.32) | 0.4 (10.07)
  Day 1; Role-emotional (n=94,93) | 46.7 (11.46) | 45.8 (11.72)
  Change at Day 28; Role-emotional (n=94,93) | 0.0 (9.49) | -1.0 (9.99)
  Day 1; Mental health (n=94,93) | 50.4 (9.14) | 49.6 (8.80)
  Change at Day 28; Mental health (n=94,93) | 2.2 (7.29) | -0.7 (8.17)

ADVERSE EVENTS:
Time Frame: From the start of open-label period until 7 days after the last dose of study medication
Arm/Group | Tramadol Hydrochloride and Acetaminophen (Open-Label) | Tramadol Hydrochloride and Acetaminophen (Double-Blind) | Placebo (Double-Blind)
Serious Adverse Events (participants affected / at risk) | 0/277 | 1/94 | 0/93
Other Adverse Events (participants affected / at risk) | 222/277 | 47/94 | 44/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tramadol Hydrochloride and Acetaminophen (Open-Label) (N=277) | Tramadol Hydrochloride and Acetaminophen (Double-Blind) (N=94) | Placebo (Double-Blind) (N=93)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tramadol Hydrochloride and Acetaminophen (Open-Label) (N=277) | Tramadol Hydrochloride and Acetaminophen (Double-Blind) (N=94) | Placebo (Double-Blind) (N=93)
Nasopharyngitis (Infections and infestations) | 6 | 5 | 17
Oral herpes (Infections and infestations) | 2 | 0 | 0
Cystitis (Infections and infestations) | 1 | 1 | 0
Sty (Infections and infestations) | 1 | 0 | 1
Upper respiratory infection (Infections and infestations) | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 1 | 0
Loss of appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 3 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Somnolence (Nervous system disorders) | 77 | 1 | 2
Dizziness (Nervous system disorders) | 45 | 3 | 0
Headache (Nervous system disorders) | 21 | 1 | 2
Attention deficit (Nervous system disorders) | 2 | 0 | 0
Dysgeusia (Nervous system disorders) | 2 | 0 | 0
Hypoesthesia (Nervous system disorders) | 2 | 0 | 0
Tremors (Nervous system disorders) | 2 | 0 | 0
Positional vertigo (Nervous system disorders) | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 2 | 0 | 0
Meniere's disease (Ear and labyrinth disorders) | 1 | 0 | 0
Rotatory vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 1 | 0 | 0
Hot flashes (Vascular disorders) | 4 | 0 | 1
Hypertension (Vascular disorders) | 2 | 0 | 0
Blushing (Vascular disorders) | 1 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 125 | 5 | 3
Vomiting (Gastrointestinal disorders) | 76 | 1 | 1
Constipation (Gastrointestinal disorders) | 52 | 3 | 0
Gastric discomfort (Gastrointestinal disorders) | 12 | 1 | 1
Upper abdominal pain (Gastrointestinal disorders) | 9 | 2 | 2
Diarrhea (Gastrointestinal disorders) | 3 | 1 | 5
Dry mouth (Gastrointestinal disorders) | 3 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 2
Stomatitis (Gastrointestinal disorders) | 2 | 0 | 1
Cheilitis (Gastrointestinal disorders) | 1 | 1 | 0
Indigestion (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0 | 1
Abnormal gastrointestinal sounds (Gastrointestinal disorders) | 1 | 0 | 0
Liver function abnormality (Hepatobiliary disorders) | 2 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 18 | 0 | 1
Excessive perspiration (Skin and subcutaneous tissue disorders) | 13 | 0 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 5 | 0 | 0
Exanthema (Skin and subcutaneous tissue disorders) | 5 | 0 | 0
Allergic pruritus (Skin and subcutaneous tissue disorders) | 5 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Ingrown nail (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Systemic pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Heat rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Leg mass (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Hematuria (Renal and urinary disorders) | 1 | 0 | 0
Urination disorder (Renal and urinary disorders) | 1 | 0 | 0
Ischuria (Renal and urinary disorders) | 1 | 0 | 0
Abnormal sensation (General disorders) | 15 | 3 | 0
Dry mouth (General disorders) | 10 | 1 | 1
Lassitude (General disorders) | 5 | 0 | 1
Asthenia (General disorders) | 1 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 0
Fever (General disorders) | 1 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 5 | 2 | 3
Blood lactate dehydrogenase increased (Investigations) | 3 | 2 | 0
γ-glutamyl transferase increased (Investigations) | 3 | 11 | 3
Blood bilirubin increased (Investigations) | 2 | 0 | 0
Blood pressure elevated (Investigations) | 2 | 1 | 0
Blood triglycerides increased (Investigations) | 2 | 4 | 0
Blood uric acid increased (Investigations) | 2 | 1 | 0
Urine glucose positive (Investigations) | 2 | 1 | 1
Urine blood positive (Investigations) | 2 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 2 | 0
Blood creatinine decreased (Investigations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0
Blood urea increased (Investigations) | 1 | 5 | 1
Neutrophil count increased (Investigations) | 1 | 0 | 0
Eosinophil fraction increased (Investigations) | 1 | 1 | 1
Neutrophil fraction increased (Investigations) | 1 | 0 | 0
Lymphocyte fraction decreased (Investigations) | 1 | 0 | 0
Urine protein positive (Investigations) | 1 | 0 | 0
Fall/tumble (Injury, poisoning and procedural complications) | 3 | 2 | 0
Traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0
Neck injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 2 | 2
Eosinophil count increased (Investigations) | 0 | 2 | 0
Blood K increased (Investigations) | 0 | 1 | 0
Hemoglobin decreased (Investigations) | 0 | 1 | 0
Lipids increased (Investigations) | 0 | 0 | 1
Liver function test abnormality (Investigations) | 0 | 1 | 0
Weight loss (Investigations) | 0 | 1 | 0
White blood cell count increased (Investigations) | 0 | 1 | 0
Platelet count increased (Investigations) | 0 | 1 | 0
Kidney function test abnormality (Investigations) | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 2
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 1
Convulsions (Nervous system disorders) | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0
Abnormal sensation in the eye (Eye disorders) | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 1
Vision impairment (Eye disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Upper respiratory inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Glossitis (Gastrointestinal disorders) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PIs is that the Sponsor can review results communications prior to public release.